CLINICAL TRIAL: NCT03442296
Title: Baltimore HEARS Study: Addressing Hearing Impairment and Social Engagement Through Community-delivered Hearing Care
Brief Title: Baltimore HEARS: Hearing Health Equity Through Accessible Research & Solutions
Acronym: HEARS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00144968; R33DC015062-03 (NIH)
Record Dates: First submitted 2018-02-06; First posted 2018-02-22 (Actual); Results first posted 2021-10-14 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-09

CONDITIONS: Age-related Hearing Impairment 1; Personal Communication
MeSH Terms: conditions — Age-Related Hearing Impairment 1; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment Group (Experimental): Immediate treatment with Baltimore HEARS intervention
  Interventions: Behavioral: Baltimore HEARS; Device: Baltimore HEARS
- Delayed Treatment Group (Placebo Comparator): 3-month delayed treatment with Baltimore HEARS intervention
  Interventions: Behavioral: Baltimore HEARS; Device: Baltimore HEARS

INTERVENTIONS:
Behavioral: Baltimore HEARS — Tailored aural rehabilitation for participant and communication partner (if applicable)
Device: Baltimore HEARS — Tailored fitting and programming of a personal sound amplifier. This will be accompanied by a component of aural rehabilitation.

SUMMARY:
Age-related hearing loss is highly prevalent and hearing health care is underutilized. The primary objective of the proposed randomized controlled trial is to investigate the efficacy of a community health worker (CHW)-delivered hearing loss intervention program. A preceding pilot study demonstrated preliminary effectiveness of the intervention program in reducing self-reported hearing handicap, and highlighted its acceptability among the target demographic. The proposed trial will now expand upon lessons learned through previous pilot studies and expand to other affordable residences for low-to-moderate income older adults in Baltimore. Primary outcome measurements will investigate intervention effects on hearing handicap, with secondary measurements investigating effects on domains such as social isolation and quality of life. This trial is a first-in-kind investigation of a novel community-based intervention that addresses hearing loss in a vulnerable, urban population.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 years or older
* English-speaking
* Aural-oral verbal communication as primary communication modality
* Post-lingual hearing loss (Audiometric pure tone averages [0.5-4kHz] in both ears >25 dB)
* Does not currently use a hearing amplification device or hearing aid
* Signed informed consent to participate in all study related activities
* Willing to regularly use listening device once provided for the remainder of their time in the study
* Hearing handicap as measured by HHIE-S score >8
* Able to follow study instructions

Exclusion Criteria:

* Individuals who do not fulfill inclusion criteria
* Evidence of ear disease or pathology requiring further medical evaluation

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-04-18 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2021-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank R Lin, MD, PhD, Principal Investigator — Johns Hopkins University; Carrie L Nieman, MD, MPH, Study Director — Johns Hopkins University
Locations (2):
- United States (2):
  - Catholic Charities, Baltimore, Maryland
  - Weinberg Senior Living Communities, Baltimore, Maryland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ventry IM, Weinstein BE. Identification of elderly people with hearing problems. ASHA. 1983 Jul;25(7):37-42. No abstract available. PMID 6626295
- [Background] Weinstein BE. Validity of a screening protocol for identifying elderly people with hearing problems. ASHA. 1986 May;28(5):41-5. No abstract available. PMID 3718608
- [Background] Tuley MR, Mulrow CD, Aguilar C, Velez R. A critical reevaluation of the Quantified Denver Scale of Communication Function. Ear Hear. 1990 Feb;11(1):56-61. doi: 10.1097/00003446-199002000-00011. PMID 2307305
- [Background] Russell D, Peplau LA, Cutrona CE. The revised UCLA Loneliness Scale: concurrent and discriminant validity evidence. J Pers Soc Psychol. 1980 Sep;39(3):472-80. doi: 10.1037//0022-3514.39.3.472. PMID 7431205
- [Background] Stewart AL, Hays RD, Ware JE Jr. The MOS short-form general health survey. Reliability and validity in a patient population. Med Care. 1988 Jul;26(7):724-35. doi: 10.1097/00005650-198807000-00007. No abstract available. PMID 3393032
- [Derived] Nieman CL, Betz J, Garcia Morales EE, Suen JJ, Trumbo J, Marrone N, Han HR, Szanton SL, Lin FR. Effect of a Community Health Worker-Delivered Personal Sound Amplification Device on Self-Perceived Communication Function in Older Adults With Hearing Loss: A Randomized Clinical Trial. JAMA. 2022 Dec 20;328(23):2324-2333. doi: 10.1001/jama.2022.21820. PMID 36538311
- [Derived] Marrone NL, Nieman CL, Coco L. Community-Based Participatory Research and Human-Centered Design Principles to Advance Hearing Health Equity. Ear Hear. 2022 Jul-Aug 01;43(Suppl 1):33S-44S. doi: 10.1097/AUD.0000000000001183. Epub 2020 Jun 13. PMID 35724253
- See also: Description of HHIE - S measure — https://consultgeri.org/try-this/general-assessment/issue-12

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study recruitment began in April 2018 and ended in October 2019. Participants were recruited from independent senior housing in Baltimore City and County and from Baltimore City senior centers and social centers.
Period: 3 Month Follow-up
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Started | 78 | 73
Completed | 73 | 70
Not Completed | 5 | 3
Not completed — Death | 3 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Obtained Hearing Aids | 0 | 1
Period: 12 Month Follow-up
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Started | 58 (15 participants in the immediate group did not start the 12month visit due to: death unrelated to study (3), loss to follow up (8), or withdrew consent (4)) | 52 (18 participants in the delayed group did not start the 12month visit due to: death unrelated to study (3), loss to follow up (5), or withdrew consent (10))
Completed | 57 | 51
Not Completed | 1 | 1
Not completed — Incomplete measurement | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Treatment Group | Delayed Treatment Group | Total
Number analyzed (Participants) | 78 | 73 | 151
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.1 (7.1) | 78.2 (8.8) | 77.1 (8)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Sex: Female | 47 | 54 | 101
  Sex: Male | 31 | 17 | 48
  Sex: NA | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Black | 40 | 25 | 65
  Race/Ethnicity: Hispanic | 1 | 2 | 3
  Race/Ethnicity: White Not Hispanic | 37 | 39 | 76
  Race/Ethnicity: Other | 0 | 7 | 7
Living Arrangement [Count of Participants; unit: Participants]
  Does not live alone | 25 | 17 | 42
  Lives Alone | 53 | 56 | 109
Education [Count of Participants; unit: Participants]
  High School or Equivalent | 20 | 22 | 42
  Less than High School | 21 | 21 | 42
  More than High School | 37 | 30 | 67
Monthly Household Income [Count of Participants; unit: Participants]
  Less than $25,000 | 48 | 48 | 96
  $25,000 to $49,999 | 16 | 16 | 32
  $50,000 to $74,999 | 7 | 4 | 11
  $75,000 to $99,999 | 2 | 2 | 4
  $100,000 to $149,999 | 0 | 1 | 1
  Don't Know | 3 | 1 | 4
  Refused | 2 | 0 | 2
  Skipped | 0 | 1 | 1
Montreal Cognitive Assessment [Mean (Standard Deviation); unit: score on a scale] — Measure was collected through a one-on-one interview with a trained data collector.
  The MoCA is a cognitive screening test designed to assist Health Professionals in the detection of mild cognitive impairment and Alzheimer's disease. Not used for diagnostic purposes. Scored from 0-30. Presented scores have been adjusted for low education. Lower scores may be interpreted as more severe cognitive impairment. Population: 1 survey missing from immediate group. 1 survey refused from immediate group
  score on a scale
    number analyzed (Participants) | 76 | 73 | 149
    (all) | 22.6 (4.4) | 23.5 (3.9) | 23 (4.2)
Speech-Frequency Pure Tone Average [Mean (Standard Deviation); unit: db HL] — Measure was collected via a portable audiometer with a trained data collector certified in hearing screening by the study audiologist and study investigator.
  Audiometric pure tone averages [0.5-4kHz] in both ears
  db HL | 41.5 (12.8) | 42.6 (11.2) | 42 (12)
Hearing Loss [Count of Participants; unit: Participants]
  Mild | 43 | 35 | 78
  Moderate to severe | 35 | 38 | 73
Prior Hearing Aid Use [Count of Participants; unit: Participants]
  No prior Hearing Aid Use | 66 | 52 | 118
  Prior Hearing Aid Use | 11 | 21 | 32
  Don't Know | 1 | 0 | 1
HHIE-S (Hearing handicap inventory for the elderly - screening) [Mean (Standard Deviation); unit: score on a scale] — Measure was collected through a one-on-one interview with a trained data collector.
  This measure is a self-reported survey on hearing handicap. Total 10 questions, up to 4 points a question. Lower scores indicate less hearing handicap.
  Scoring:
  0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap Population: 2 incomplete surveys from the immediate group
  score on a scale
    number analyzed (Participants) | 76 | 73 | 149
    (all) | 21.7 (9.4) | 20.1 (10.1) | 21 (9.7)
UCLA Loneliness Scale [Mean (Standard Deviation); unit: score on a scale] — Measure was collected via a one-on-one interview conducted by a trained data collector.
  20-item Likert-type scale. Total score is sum of the 20 items, scores range from 20 to 80. Lower values equate to lower levels of loneliness and higher values equate to higher levels of loneliness.
  Score ranges:
  20-34 - Low degree of loneliness 35-49 - Moderate degree of loneliness 50-64 - Moderately high degree of loneliness 65-80 - High degree of loneliness Population: 5 incomplete surveys not included (3 immediate, 2 delayed)
  score on a scale
    number analyzed (Participants) | 75 | 71 | 146
    (all) | 23.3 (10) | 20.6 (9.2) | 22 (9.7)
Patient Health Questionnaire - Depression Score (PHQ-9) [Mean (Standard Deviation); unit: score on a scale] — Measure collected via one-on-one interview conducted by trained data collectors.
  Total of 9 questions, scored from 0 to 3. The score from each question are summed to a total score, which can range from 0 to 27.
  Interpretation of Total Score Total Score Depression Severity 0 No depression 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression Population: 8 incomplete surveys not included (3 immediate, 5 delayed)
  score on a scale
    number analyzed (Participants) | 75 | 68 | 143
    (all) | 6 (4.5) | 5.9 (4.5) | 6 (4.5)
Cohen Social Network Index (SNI): Network Diversity [Mean (Standard Deviation); unit: number of roles] — Measure was collected through a one-on-one interview with a trained data collector.
  This measure is the number of types of high contact roles a participant self reports to have interacted with in the past 2 weeks (family, friends, etc.). Maximum count of 12. Population: 8 incomplete measures not included (5 immediate, 3 delayed)
  number of roles
    number analyzed (Participants) | 73 | 70 | 143
    (all) | 4.8 (1.9) | 4.9 (1.7) | 4.8 (1.8)
Cohen Social Network Index (SNI): Social Network Size [Median (Inter-Quartile Range); unit: number of people] — Measure was collected through a one-on-one interview with a trained data collector.
  This measure is a self-reported number of individuals in a high contact role that a participant has interacted with in the past 2 weeks. Maximum number of 103. Population: 8 incomplete measures not included (5 immediate, 3 delayed)
  number of people
    number analyzed (Participants) | 73 | 70 | 143
    (all) | 17 [11 to 22] | 15.5 [10 to 21] | 16 [10 to 22]
12-Item Short Form Survey (SF-12): Mental Component Score [Mean (Standard Deviation); unit: score on a scale] — The 12-Item Short Form Survey (SF-12) was collected through a one-on-one interview with a trained data collector.
  The 12-Item Short Form Survey (SF-12) measures the construct of self-reported health-related quality of life. Here we report the mental component which relates to mental health functioning. Score ranges from 0-100 with higher scores indicating better mental health functioning. Population: 6 incomplete measures not included (3 immediate, 3 delayed)
  score on a scale
    number analyzed (Participants) | 75 | 70 | 145
    (all) | 48.5 (10.1) | 49.4 (9.9) | 49 (10)
12-Item Short Form Survey (SF-12) Physical Component Score [Mean (Standard Deviation); unit: score on a scale] — The 12-Item Short Form Survey (SF-12) was collected through a one-on-one interview with a trained data collector.
  The 12-Item Short Form Survey (SF-12) measures the construct of self-reported health-related quality of life. Here we report the physical component which relates to physical health functioning. Score ranges from 0-100 with higher scores indicating better physical health functioning. Population: 6 incomplete measures not included (3 immediate, 3 delayed)
  score on a scale
    number analyzed (Participants) | 75 | 70 | 145
    (all) | 39 (11) | 39.4 (11.1) | 39.2 (11)
Rapid Estimate of Adult Literacy in Medicine-Short Form (REALM-SF) [Mean (Standard Deviation); unit: score on a scale] — Measure was collected through a one-on-one interview with a trained data collector.
  This measure is 7-item word recognition test to provide a valid quick assessment of participant health literacy. Score ranges from 0 to 7, higher scores meaning higher health literacy and lower scores meaning lower health literacy. Population: 1 incomplete measure not included from immediate group
  score on a scale
    number analyzed (Participants) | 77 | 73 | 150
    (all) | 6.1 (1.7) | 6.1 (1.8) | 6.1 (1.8)
Adapted from Attitudes Towards Computers Questionnaire (ATCQ): Computer Self Efficacy [Mean (Standard Deviation); unit: score on a scale] — Measure was collected via a one- on-one interview conducted by a trained data collector. 5 question survey of self-reported computer self-efficacy on a 5-point Likert scale. Score range: 0 - 25 points. Higher score indicates higher self-efficacy.
  score on a scale | 19.3 (3.9) | 19.1 (4.6) | 19.2 (4.3)
Adapted from Attitudes Towards Computers Questionnaire (ATCQ): Listening Device Interest [Mean (Standard Deviation); unit: units on a scale] — Measure was collected via a one- on-one interview conducted by a trained data collector. 5 question survey of self-reported listening device interest on a 5-point Likert scale. Score range: 0 - 25 points. Higher score indicate higher interest.
  units on a scale | 13.9 (1.8) | 14.3 (1.8) | 14.1 (1.8)
Adapted from Attitudes Towards Computers Questionnaire (ATCQ): Listening Device Self Efficacy [Mean (Standard Deviation); unit: units on a scale] — Measure was collected via a one- on-one interview conducted by a trained data collector. 5 question survey of self-reported listening device self efficacy on a 5-point Likert scale. Score range: 0-25 points. Higher score indicate higher self efficacy. Population: 3 incomplete measures not included (1 immedaite, 2 delayed)
  units on a scale
    number analyzed (Participants) | 77 | 71 | 148
    (all) | 21.7 (2.3) | 20.9 (3.1) | 21.3 (2.7)
Own Smartphone [Count of Participants; unit: Participants]
  Doesn't own smartphone | 36 | 32 | 68
  Owns smartphone | 42 | 40 | 82
  NA | 0 | 1 | 1
Used Computer within past month [Count of Participants; unit: Participants]
  "I do not have or use a computer" | 38 | 38 | 76
  "I have or use a computer but I do not go on the internet" | 9 | 6 | 15
  "I have or use a computer and I used the internet" | 31 | 29 | 60
Used text or email within the past month [Count of Participants; unit: Participants]
  Most days | 27 | 24 | 51
  Some days | 8 | 13 | 21
  Rarely | 10 | 10 | 20
  Not within the past month | 33 | 26 | 59
Adapted from Listening Self-Efficacy Questionnaire (LSEQ): Total Score [Mean (Standard Deviation); unit: score on a scale] — Measure was collected through a one-on-one interview with a trained data collector. 5 question survey on self reported self-efficacy in different listening situations on a 0-10 scale. A higher score means higher self-efficacy. Maximum score of 50. Population: 2 incomplete baseline measures in the delayed group
  score on a scale
    number analyzed (Participants) | 78 | 71 | 149
    (all) | 28.9 (10.3) | 28.9 (9.1) | 28.9 (9.7)
Adapted from Listening Self-Efficacy Questionnaire (LSEQ): Complex Listening Self- Efficacy [Mean (Standard Deviation); unit: score on a scale] — Measure was collected through a one-on-one interview with a trained data collector. This measure is the combined score of two questions where a participant self-reported their listening self efficacy on a 0-10 scale in complex listening situations. Participants answer with a higher number the more confident they are in the presented situation. Score ranges from 0 to 20. Population: 1 incomplete baseline measure in the delayed group
  score on a scale
    number analyzed (Participants) | 78 | 72 | 150
    (all) | 7.7 (4.9) | 7.3 (4.7) | 7.6 (4.8)
Adapted from Listening Self-Efficacy Questionnaire (LSEQ): Directed Listening Self-Efficacy [Mean (Standard Deviation); unit: score on a scale] — Measure was collected through a one-on-one interview with a trained data collector. This measure is the combined score of two questions where a participant self-reported their listening self efficacy on a 0-10 scale in directed listening situations. Participants answer with a higher number the more confident they are in the presented situation. Score ranges from 0 to 20. Population: 2 incomplete baseline measures in the delayed group
  score on a scale
    number analyzed (Participants) | 78 | 71 | 149
    (all) | 13.7 (4.5) | 13.8 (4) | 13.8 (4.2)
Adapted from Listening Self-Efficacy Questionnaire (LSEQ): Dialog in Quiet Listening Self-Efficacy [Mean (Standard Deviation); unit: score on a scale] — Measure was collected through a one-on-one interview with a trained data collector. This measure has the participant self report their listening self efficacy on a 0-10 scale in a dialog in quiet listening situation. Participants answer with a higher number the more confident they are in the presented situation. Maximum possible score is 10. Population: 1 incomplete baseline measure in delayed group
  score on a scale
    number analyzed (Participants) | 78 | 72 | 150
    (all) | 7.4 (2.5) | 7.7 (2.2) | 7.6 (2.4)
Hearing Knowledge [Mean (Standard Deviation); unit: score on a scale] — Measure was collected through a one-on-one interview with a trained data collector . This 5 question measure asks participants about their hearing knowledge. Score ranges from 0 to 5. Higher score indicates greater hearing knowledge. Population: 9 incomplete baseline measures (5 immediate, 4 delayed)
  score on a scale
    number analyzed (Participants) | 73 | 69 | 142
    (all) | 3.3 (1.5) | 3.4 (1.7) | 3.4 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hearing Handicap Inventory for the Elderly (HHIE-S)
Description: Measure was collected through a one-on-one interview with a trained data collector. Higher scores indicate increased hearing handicap.
  Scoring:
  0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap
  Change from baseline is reported. An increase in the score from baseline (a positive number) indicates a worsening in hearing handicap.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 4 incomplete baseline measures (2 immediate, 2 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  3 incomplete 3 month measures from immediate group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 68 | 68
score on a scale | -13.2 (10.3) | .06 (7.1)

2. Secondary Outcome: Change From Baseline in Revised UCLA Loneliness Scale
Description: Measure was collected via a one-on-one interview conducted by a trained data collector.
  Score is the sum of 20-item self-reported measure. Scores range from 20 to 80.
  Score ranges:
  20-34 - Low degree of loneliness 35-49 - Moderate degree of loneliness 50-64 - Moderately high degree of loneliness 65-80 - High degree of loneliness.
  Change from baseline is reported. An increase in the score from baseline (a positive number) indicates a worsening in degree of loneliness.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 5 incomplete baseline measures (3 immediate, 2 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  16 incomplete 3 month measures (11 immediate, 5 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 59 | 63
score on a scale | -2.8 (8.7) | -0.6 (7)

3. Secondary Outcome: Change From Baseline in Self-reported Depression in Patient Health Questionnaire (PHQ-9)
Description: Measure collected via one-on-one interview conducted by trained data collectors.
  Total of 9 questions, scored from 0 to 3. The score from each question are summed to a total score, which can range from 0 to 27.
  Interpretation of Total Score Total Score Depression Severity 0 No depression 1-4 Minimal depression 5-9 Mild depression 10-14 Moderate depression 15-19 Moderately severe depression 20-27 Severe depression.
  Change from baseline is reported. An increase in the score from baseline (a positive number) indicates a worsening in depression severity.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 8 incomplete baseline measures (3 immediate, 5 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  11 incomplete 3 month measures (9 immediate, 2 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 61 | 63
score on a scale | -1 (4.3) | -0.2 (4)

4. Secondary Outcome: Change From Baseline in Short Form-12 (SF-12) Mental Component Score
Description: The 12-Item Short Form Survey (SF-12) was collected through a one-on-one interview with a trained data collector.
  The 12-Item Short Form Survey (SF-12) measures the construct of self-reported health-related quality of life. Here we report the mental component which relates to mental health functioning. Score ranges from 0-100 with higher scores indicating better mental health functioning.
  Change from baseline is reported. An increase in the score from baseline (a positive number) indicates a better health state.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 6 incomplete baseline measures (3 immediate, 3 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  12 incomplete 3 month measures (11 immediate, 1 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 59 | 66
score on a scale | 1.1 (11.2) | -1.4 (10)

5. Secondary Outcome: Change From Baseline in Short Form -12 (SF-12) Physical Component Score
Description: The 12-Item Short Form Survey (SF-12) was collected through a one-on-one interview with a trained data collector.
  The 12-Item Short Form Survey (SF-12) measures the construct of self-reported health-related quality of life. Here we report the physical component which relates to physical health functioning. Score ranges from 0-100 with higher scores indicating better physical health functioning.
  Change from baseline is reported. An increase in the score from baseline (a positive number) indicates a better health state.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 59 | 66
score on a scale | 4.4 (10.4) | -0.4 (10.1)

6. Secondary Outcome: Change From Baseline in Cohen Social Network Index (SNI): Network Diversity
Description: Change from baseline in total number of high contact roles the participant interacts with at least every 2 weeks (such as family, friends, work). Maximum of 12 roles included on the measure. An increase in the score from baseline (a positive number) indicates a more diverse network.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 5 incomplete measures at baseline (3 immediate, 2 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  17 incomplete 3 month measures (12 immediate, 5 delayed)
Measure: Mean (Standard Deviation); unit: number of roles
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 58 | 63
number of roles | 0.3 (1.2) | -0.0 (1.2)

7. Secondary Outcome: Change From Baseline in Cohen Social Network Index (SNI): Social Network Size
Description: Change from baseline in total number of individuals in high contact roles the participant interacts with at least every 2 weeks (such as family, friends, work). .An increase in the number of individuals from baseline (a positive number) indicates an increase in their social network size.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 5 incomplete baseline measures (3 immediate, 2 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  17 incomplete 3 month measures (12 immediate, 5 delayed)
Measure: Mean (Standard Deviation); unit: number of individuals
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 58 | 63
number of individuals | 1.8 (10.5) | 1.0 (7.2)

8. Secondary Outcome: Change From Baseline in Valuation of Life
Description: This self-reported 13 question measure asks the participant how much they agree or disagree on a 5 point Likert scale when asked a statement about the meaning of life and personal goals. Score ranges from 0 to 65. Higher score means higher value of life.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher value of life.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 7 incomplete baseline measures (3 immediate, 4 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  11 incomplete 3 month measures (10 immediate, 1 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 60 | 65
score on a scale | 0.1 (6.9) | -0.6 (5.1)

9. Secondary Outcome: Change From Baseline in Adapted From Attitudes Towards Computers Questionnaire (ATCQ): Computer Self-Efficacy
Description: A 5 question measure surveying self-reported self-efficacy of computer use on a 5 point Likert scale. Score ranges from 0 to 25.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher self-efficacy.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  12 incomplete 3 month measures (11 immediate, 1 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 62 | 69
score on a scale | -0.5 (3.8) | 0 (3.2)

10. Secondary Outcome: Change From Baseline in Adapted From Attitudes Towards Computers Questionnaire (ATCQ): Device Self-Efficacy
Description: A 5 question measure surveying self-reported device self-efficacy on a 5 point Likert scale. Score ranges from 0 to 25.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher self-efficacy.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 3 incomplete baseline measures (1 immediate, 2 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  10 incomplete 3 month measures from immediate group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 62 | 68
score on a scale | -0.6 (3.8) | -0.1 (3.6)

11. Secondary Outcome: Change From Baseline in Adapted From Attitudes Towards Computers Questionnaire (ATCQ): Listening Device Interest
Description: A 5 question measure surveying self-reported self-efficacy of listening device interest on a 5 point Likert scale. Score ranges from 0 to 25.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher self-efficacy.
Time Frame: Baseline and 3 months post-intervention (Immediate Group) or 3 months post-baseline (Delayed Group)
Population: 1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  10 incomplete 3 month measures in immediate group
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 63 | 70
score on a scale | 0.7 (2.3) | -0.4 (2.5)

12. Secondary Outcome: Change From Baseline in Adapted From Listening Self-Efficacy Questionnaire (LSEQ): Total Score
Description: This 5 question survey measures listening self efficacy on a 0-10 scale in different situations such as being able to understand a conversation in a quiet room to a crowded restaurant. Participants answer with a higher number the more confident they are in the presented situation. Maximum possible score is 50.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher self-efficacy.
Time Frame: Baseline and 3 month post-intervention (immediate group) or 3 month post-baseline (delayed group)
Population: 2 incomplete baseline measures (2 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  12 incomplete 3 month measures (12 immediate)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 61 | 68
score on a scale | 10.8 (11.3) | -0.7 (8.1)

13. Secondary Outcome: Change From Baseline in Adapted From Listening Self-Efficacy Questionnaire (LSEQ): Complex Listening
Description: This measure is the combined score of two questions where a participant self-reported their listening self efficacy on a 0-10 scale in complex listening situations. Participants answer with a higher number the more confident they are in the presented situation. Score ranges from 0 to 20.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher self-efficacy.
Time Frame: Baseline and 3 month post-intervention (immediate group) or 3 month post-baseline (delayed group)
Population: 1 incomplete baseline measures (1 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  12 incomplete 3 month measures (12 immediate)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 61 | 69
score on a scale | 5.1 (5.7) | -0.1 (4.3)

14. Secondary Outcome: Change From Baseline in Adapted From Listening Self-Efficacy Questionnaire (LSEQ): Directed Listening
Description: as for outcome 13
Time Frame: Baseline and 3 month post-intervention (immediate group) or 3 month post-baseline (delayed group)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 61 | 68
score on a scale | 4.2 (5.1) | -0.1 (4.5)

15. Secondary Outcome: Change From Baseline in Adapted From Listening Self-Efficacy Questionnaire (LSEQ): Dialog in Quiet
Description: This measure is a participant's self-reported listening self efficacy on a 0-10 score scale in a dialog in quiet listening situation. Participants answer with a higher number the more confident they are in the presented situation. Maximum possible score is 10.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher self-efficacy.
Time Frame: Baseline and 3 month post-intervention (immediate group) or 3 month post-baseline (delayed group)
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 61 | 69
score on a scale | 1.5 (2.7) | -0.6 (2.8)

16. Secondary Outcome: Change From Baseline in Hearing Knowledge
Description: This 5 question measure asks participants about their hearing knowledge based on the information presented in the intervention. The score ranges from 0 to 5.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates more hearing knowledge.
Time Frame: Baseline and 3 month post-intervention (immediate group) or 3 month post-baseline (delayed group)
Population: 9 incomplete baseline measures (5 immediate, 4 delayed)
  1 obtained hearing aids (1 delayed)
  1 withdrew consent (1 immediate)
  4 non-study related deaths (3 immediate, 1 delayed)
  2 lost to follow up (1 immediate, 1 delayed)
  14 incomplete 3 month measures (12 immediate, 2 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 56 | 64
score on a scale | 0.2 (1.6) | -0.4 (1.5)

17. Secondary Outcome: Change From Baseline in Hearing Handicap Inventory for the Elderly (HHIE-S)
Description: Measure was collected through a one-on-one interview with a trained data collector. Higher scores indicate increased hearing handicap.
  Scoring:
  0-8 suggests no hearing handicap 10-24 suggests mild-moderate hearing handicap 26-40 suggests significant hearing handicap.
  Change from baseline is reported. An increase in the score from baseline (a positive number) indicates a worsening in hearing handicap.
Time Frame: Baseline and 12 months post-intervention
Population: 4 incomplete baseline measure (2 immediate, 2 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  8 incomplete 12 month measures (6 immediate, 3 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 55 | 50
score on a scale | -10.3 (11) | -8.2 (13.4)

18. Secondary Outcome: Change From Baseline in Revised UCLA Loneliness Scale
Description: as for outcome 2
Time Frame: Baseline and 12 months post-intervention
Population: 5 incomplete baseline measure (3 immediate, 2 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  30 incomplete 12 month measures (19 immediate, 11 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 41 | 42
score on a scale | -1.3 (6.8) | -1.9 (9.0)

19. Secondary Outcome: Change From Baseline in Self-reported Depression in Patient Health Questionnaire (PHQ-9)
Description: as for outcome 3
Time Frame: Baseline and 12 months post-intervention
Population: 8 missing at baseline (3 immediate, 5 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  22 Incomplete 12 month measures (8 immediate, 14 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 49 | 39
score on a scale | -0.3 (3.3) | -1.1 (4.5)

20. Secondary Outcome: Change From Baseline in Short Form -12 (SF-12) Mental Component Score
Description: as for outcome 4
Time Frame: Baseline and 12 months post-intervention
Population: 6 incomplete at baseline (3 immediate, 3 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  27 incomplete 12 month measures (12 immediate, 15 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 48 | 37
score on a scale | 0.5 (9.9) | 0.7 (13.0)

21. Secondary Outcome: Change From Baseline in Short Form -12 (SF-12) Physical Component Score
Description: as for outcome 5
Time Frame: Baseline and 12 months post-intervention
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 48 | 37
score on a scale | 1.0 (9.3) | 1.7 (11.4)

22. Secondary Outcome: Change From Baseline in Cohen (Social Network Index) SNI: Network Diversity
Description: Change from baseline in total number of high contact roles the participant interacts with at least every 2 weeks (such as family, friends, work). Maximum of 12 roles included on the measure. An increase in the number of roles from baseline (a positive number) indicates a more diverse network.
Time Frame: Baseline and 12 months post-intervention
Population: 5 incomplete at baseline (3 immediate, 2 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  27 incomplete 12 month measures (15 immediate, 12 delayed)
Measure: Mean (Standard Deviation); unit: contact roles
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 45 | 41
contact roles | -0.1 (1.0) | -0.2 (1.3)

23. Secondary Outcome: Change From Baseline in Cohen Social Network Index (SNI): Social Network Size
Description: as for outcome 7
Time Frame: Baseline and 12 months post-intervention
Population: 5 incomplete at baseline (3 immediate, 2 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  27 incomplete at 12 month (15 immediate, 12 delayed)
Measure: Mean (Standard Deviation); unit: individuals
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 45 | 41
individuals | -1.5 (12.4) | -3.7 (10.4)

24. Secondary Outcome: Change From Baseline in Valuation of Life
Description: as for outcome 8
Time Frame: Baseline and 12 months post-intervention
Population: 7 incomplete baseline (3 immediate, 4 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  25 incomplete 12 month measures (14 immediate, 11 delay)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 46 | 40
score on a scale | -1.9 (6.6) | -1.0 (7.6)

25. Secondary Outcome: Change From Baseline in Adapted From Attitudes Towards Computers Questionnaire (ATCQ): Device Self-Efficacy
Description: as for outcome 10
Time Frame: Baseline and 12 months post-intervention
Population: 3 incomplete at baseline (1 immediate, 2 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  28 incomplete 12 month measures (14 immediate, 14 delay)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 48 | 39
score on a scale | -0.6 (3.5) | -0.4 (3.0)

26. Secondary Outcome: Change From Baseline in Adapted From Attitudes Towards Computers Questionnaire (ATCQ): Computer Self-Efficacy
Description: as for outcome 9
Time Frame: Baseline and 12 months post-intervention
Population: 0 incomplete baseline (0 immediate, 0 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  28 incomplete 12 month measures (14 immediate, 14 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 49 | 41
score on a scale | 0.3 (3.9) | 0.2 (2.9)

27. Secondary Outcome: Change From Baseline in Adapted From Attitudes Towards Computers Questionnaire (ATCQ): Listening Device Interest
Description: as for outcome 11
Time Frame: Baseline and 12 months post-intervention
Population: 0 incomplete at baseline (0)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  28 incomplete 12 month measures (14 immediate, 14 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 49 | 41
score on a scale | 0.9 (2.2) | 0.1 (2.0)

28. Secondary Outcome: Change From Baseline in Adapted From Listening Self-Efficacy Questionnaire (LSEQ): Total Score
Description: as for outcome 12
Time Frame: Baseline and 12 months post-intervention
Population: 2 incomplete at baseline (0 immediate, 2 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  28 incomplete 12 month measures (14 immediate, 14 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 49 | 39
score on a scale | 8.3 (9.3) | 8.2 (10.7)

29. Secondary Outcome: Change From Baseline in Adapted From Listening Self-Efficacy Questionnaire (LSEQ): Complex Listening
Description: as for outcome 13
Time Frame: Baseline and 12 months post-intervention
Population: 1 incomplete at baseline (0 immediate, 1 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  28 incomplete 12 month measures (14 immediate, 14 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 49 | 40
score on a scale | 4.0 (5.6) | 4.8 (5.3)

30. Secondary Outcome: Change From Baseline in Adapted From Listening Self-Efficacy Questionnaire (LSEQ): Directed Listening
Description: This measure is the combined score of two questions where a participant self-reported their listening self efficacy on a 0-10 scale in directed listening situations. Participants answer with a higher number the more confident they are in the presented situation. Score ranges from 0 to 20.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher self-efficacy.
Time Frame: Baseline and 12 months post-intervention
Population: 2 incomplete baseline measure (0 immediate, 2 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  28 incomplete 12 month measures (14 immediate, 14 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 49 | 39
score on a scale | 2.8 (3.8) | 2.5 (4.5)

31. Secondary Outcome: Change From Baseline in Adapted From Listening Self-Efficacy Questionnaire (LSEQ): Dialog in Quiet
Description: This measure is a participant's self-reported listening self efficacy on a 0-10 scale in a directed listening situation. Participants answer with a higher number the more confident they are in the presented situation. Maximum possible score is 10.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates a higher self-efficacy.
Time Frame: Baseline and 12 months post-intervention
Population: 1 incomplete at baseline (0 immediate, 1 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  29 incomplete 12 month measures (14 immediate, 15 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 49 | 39
score on a scale | 1.5 (1.9) | 0.8 (2.8)

32. Secondary Outcome: Change From Baseline in Hearing Knowledge
Description: This 5 question measure asks participants about their hearing knowledge based on the information presented in the intervention. Score ranges from 0 to 5.
  Change from baseline score is reported. An increase in the score from baseline (a positive number) indicates more hearing knowledge.
Time Frame: Baseline and 12 months post-intervention
Population: 9 incomplete at baseline (5 immediate, 4 delayed)
  14 withdrew consent (4 immediate, 10 delayed)
  6 non-study related deaths (3 immediate, 3 delayed)
  13 lost to follow up (8 immediate, 5 delayed)
  27 incomplete 12 month measures (12 immediate, 15 delayed)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
Number analyzed (Participants) | 46 | 36
score on a scale | 0.2 (1.7) | 0.0 (1.7)

ADVERSE EVENTS:
Time Frame: Adverse event data for each participant is collected from Screening to 12 Month Post-Intervention Visit (up to 2 years)
Arm/Group | Immediate Treatment Group | Delayed Treatment Group
All-Cause Mortality (participants affected / at risk) | 6/78 | 4/73
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/73
Other Adverse Events (participants affected / at risk) | 0/78 | 0/73

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/96/NCT03442296/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT03442296/SAP_001.pdf